CLINICAL TRIAL: NCT04867759
Title: Uterine Natural Killer (uNK) Cell Expression in Patients With Repeated ICSI Failures: A Multicenter Cohort Study
Acronym: UNK
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Collaborators: Mansoura University (Other); Benha University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Assistant professor, Tanta University
Other Study IDs: uNK in ICSI failure
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Repeated Implantation Failure; ICSI Failure; uNatural Killer Cells

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endometrial biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: On outpatient basis, we will take a uterine sample on mid-luteal phase day 21 by Novac curette or pipelle aspirator. Samples of endometrium will be kept in formaline solution and will be sent to National Institute of research and medical sceinces at Alexandria University to be tested for uNK Cells CD56.
  Interventions: Procedure: Endometrial Biopsy
- Control group: On outpatient basis, we will take a uterine sample on mid-luteal phase day 21 by Novac curette or pipelle aspirator. Samples of endometrium will be kept in formaline solution and will be sent to National Institute of research and medical sceinces at Alexandria University to be tested for uNK Cells CD56.
  Interventions: Procedure: Endometrial Biopsy

INTERVENTIONS:
Procedure: Endometrial Biopsy — On outpatient basis, we will take a uterine sample on mid-luteal phase day 21 by Novac curette or pipelle aspirator. Samples of endometrium will be kept in formaline solution and will be sent to National Institute of research and medical sceinces at Alexandria University to be tested for uNK Cells CD56.

SUMMARY:
uterine NK (uNK) cells are characterized by a high expression of CD56 (CD56brihgt), lack of CD16 expression, high secretion of cytokines and rather low cytotoxic activity. It has been shown that uNK cells increase in number during the late secretory phase and during early pregnancy. This study was designed to assess the possible role of uNK cells in repeated ICSI failure.

DETAILED DESCRIPTION:
For occurrence of the "window of implantation", the endometrium must proliferate, increase in thickness, then, after ovulation, adequately respond to progesterone, and become receptive. Ultrasound examination of the thickness and appearance of the endometrium is an easily performed means of assessing morphological changes occurring in the endometrium during the follicular phase, and is thus used as a measure to predict successful implantation. Indeed, several studies have reported a strong association between endometrial thickness and successful implantation. However, others failed to confirm such an association. The minimal adequate endometrial thickness for successful implantation, as measured in the late proliferative phase, varies between studies, with a range of 6-8 mm. However, although rare, some investigators have reported successful implantation in an endometrium of no more than 5 mm thickness.

Uterine NK cell testing can only be done via an endometrial biopsy. Uterine natural killer cells never come into direct contact with the fetal cells-they only have direct access to placental cells.The biopsy is performed on day 21 of your menstrual cycle, when the NK cell count is at its highest. The procedure is done at outpatient clinics and results take about two weeks to receive. If your NK cell activity reading is greater than 14 % on day 21 biopsy, then diagnosed with high levels of NK cell activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IVF/ICSI failures more than 2 times
* Age 20-40 years

Exclusion Criteria:

* prior uterine surgery
* immunological disease
* previous testing to uNK cells

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Patients with repeated implantation faikure
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Level of uNK cells | 4 months
  Measurement of level of uNK cells by flowcytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Adel Elgergawy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
On valuable request
Supporting Information: Study Protocol
Time Frame: 3 months